CLINICAL TRIAL: NCT05188898
Title: Treatment of Intraosseous Periodontal Pockets by Non-surgical Therapy With Micro-instruments and Application of Hyaluronic Acid. A Randomized-controlled Clinical Trial
Brief Title: Treatment of Intraosseous Periodontal Defects With Hyaluronic Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Luca Ramaglia, Clinical Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 141/21
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Periodontal Bone Loss; Periodontal Pocket
Keywords: Hyaluronic Acid; Periodontal therapy; Periodontal Bone Loss; Intraosseous Bone Defect
MeSH Terms: conditions — Alveolar Bone Loss; Periodontal Pocket | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: The study will be designed as a double-arm randomized controlled clinical trial. The intraosseous defects of subjects allocated in HA group will be treated with MINSD and application of hyaluronic acid, while in No-HA Group only MINSD will be performed. The null hypothesis of no statistically significant differences between the two modalities for the treatment of intraosseous defects will be tested.
Who Masked: Participant
Masking Description: Only patients will be unaware of the type of treatment performed, with prior written informed consent. So, they will be divided in the two groups of study after a process of randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic acid Group (Experimental): Hyaluronic acid gel will be applied in intraosseous periodontal defects, after Minimally Invasive Non Surgical Debridement (MINSD)
  Interventions: Other: MINSD and Hyaluronic acid
- No-hyaluronic acid Group (Active Comparator): Only Minimally Invasive Non Surgical Debridement (MINSD) will be performed
  Interventions: Other: MINSD

INTERVENTIONS:
Other: MINSD and Hyaluronic acid — After local anesthesia, MINSD will be performed using an ultrasonic scaler with fine tips and micro-curette; then, a hyaluronic acid-based gel will be applied to the intraosseous periodontal pockets.
  Arms: Hyaluronic acid Group
Other: MINSD — Only subgingival mechanical debridement (MINSD) will be performed with an ultrasonic scaler with fine tips and micro-curette.
  Arms: No-hyaluronic acid Group

SUMMARY:
The aim of the present investigation will be evaluate the healing of periodontal intraosseous defects following Minimally Invasive Non Surgical Debridement (MINSD) and application of a hyaluronic acid-based gel, compared to MINSD alone.

A total of 22 patients will be enrolled, selected by inclusion and exclusion criteria and randomly divided in two groups: hyaluronic acid group (HA) and no-hyaluronic acid group (No-HA).

DETAILED DESCRIPTION:
The objective of the study will be compare the healing of periodontal intraosseous defects following treatment with Minimally Invasive Non Surgical Debridement (MINSD) and application of hyaluronic acid (HA) compared to MINSD alone.

Twenty-two patients with intraosseous periodontal defects will be randomly assigned to treatment with MINSD and application of a hyaluronic acid-based gel (HA Group) or MINSD alone (No-HA Group).

Primary outcome will be "Probing Depth" (PD), while the secondary outcomes will be "Clinical Attachment Level" (CAL) gain, "Gingival Recession" (GR) and "Radiographic Defect Angle" (RDA).

After local anesthesia, in HA group MINSD will be performed using an ultrasonic scaler with fine tips and micro-curette; then, a hyaluronic acid-based gel will be applied to the intraosseous periodontal pockets.

In the No-HA group, only subgingival mechanical debridement (MINSD) will be performed with an ultrasonic scaler with fine tips and micro-curette.

Finally, a polishing paste will be applied to the supra-gingival level in both groups using a rubber cup. Patients of both groups will be recalled every month for professional oral hygiene and, after 6 months, all measurements will be repeated and the final evaluation will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with periodontitis;
* Age ≥ 18 years old;
* Presence of at least 10 teeth per arch;
* Presence of at least two teeth with Probing Depth (PD) ≥ 5 mm per quadrant;
* Presence of at least one intraosseous pocket;
* Single-rooted and multi-rooted teeth.

Exclusion Criteria:

* Patients with systemic diseases;
* Prolonged antibiotic or anti-inflammatory treatment within 4 weeks prior to periodontal therapy;
* Pregnant or lactating;
* Tobacco smokers (≥ 10 cigarettes per day);
* Multi-rooted teeth with furcation involvement;
* Third molars.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Change of Probing Depth (PD) (millimeters) | baseline and 6 months after periodontal therapy
  Distance from the gingival margin to the bottom of the pocket

SECONDARY OUTCOMES:
Change of Clinical Attachment Level (CAL) gain (millimeters) | baseline and 6 months after periodontal therapy
  Distance from the Cement Enamel Junction (CEJ) to the bottom of the pocket
Change of Gingival Recession (GR) (millimeters) | baseline and 6 months after periodontal therapy
  Distance from gingival margin to the cementoenamel junction
Change of Radiographic Defect Angle (RDA) (grade °) | baseline and 6 months after periodontal therapy
  Radiographic intraosseous angle

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iorio-Siciliano V, Blasi A, Mauriello L, Salvi GE, Ramaglia L, Sculean A. Non-Surgical Treatment of Moderate Periodontal Intrabony Defects With Adjunctive Cross-Linked Hyaluronic Acid: A Single-Blinded Randomized Controlled Clinical Trial. J Clin Periodontol. 2025 Feb;52(2):310-322. doi: 10.1111/jcpe.14078. Epub 2024 Oct 14. PMID 39402910